CLINICAL TRIAL: NCT03222323
Title: Does Perineural Dexmedetomidine Prolong the Duration of an Ulnar Nerve Block When Controlling for Possible Systemic Effects?
Brief Title: Perineural Dexmedetomidine for Ulnar Nerve Block.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Jakob Hessel Andersen, Anesthesiologist, Staff Specialist, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REG-158-2016; 2016-004883-20 (EudraCT Number)
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Healthy
Keywords: volunteers
MeSH Terms: interventions — Dexmedetomidine; Ropivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The participants will attend two trial days and receive two treatments on each trial days
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Perineural dexmedetomidine (Experimental): Ulnar nerve block 4ml ropivacaine 5mg/ml + 1ml 100ug/ml dexmedetomidine perineurally
  Interventions: Drug: Dexmedetomidine perineurally; Drug: Ropivacaine 5mg/ml
- Systemic dexmedetomidine (Active Comparator): Ulnar nerve block 4ml ropivacaine 5mg/ml + 1ml isotonic saline (placebo) perineurally + 100ug dexmedetomidine systemically (absorbed and redistributed from the opposite ulnar nerve block)
  Interventions: Drug: Ropivacaine 5mg/ml; Drug: Dexmedetomidine systemically; Drug: Isotonic saline
- Placebo (Placebo Comparator): Ulnar nerve block 4ml ropivacaine 5mg/ml + 1ml isotonic saline (placebo) perineurally
  Interventions: Drug: Ropivacaine 5mg/ml; Drug: Isotonic saline
- High dose Ropivacaine (Active Comparator): Ulnar nerve block 4ml ropivacaine 7.5mg/ml + 1ml isotonic saline (placebo) perineurally
  Interventions: Drug: Ropivacaine 7.5mg/ml; Drug: Isotonic saline

INTERVENTIONS:
Drug: Dexmedetomidine perineurally — Dexmedetomidine is added perineurally on one side and will influence the nerve block perineurally on this side. Dexmedetomidine is also absorbed and redistributed systemically and will influence the opposite ulnar nerve block systemically.
  Other Names: Dexdor
  Arms: Perineural dexmedetomidine
Drug: Ropivacaine 5mg/ml — Ropivacaine is used in 5mg/ml in the perineural, systemic and placebo nerve blocks.
  Other Names: Naropine
  Arms: Perineural dexmedetomidine; Placebo; Systemic dexmedetomidine
Drug: Ropivacaine 7.5mg/ml — In the high dose ropivacaine group a ropivacaine concentration of 7.5mg/ml is used.
  Other Names: Naropine
  Arms: High dose Ropivacaine
Drug: Dexmedetomidine systemically — Dexmedetomidine administered perineurally on one side is absorbed and redistributed systemically and will influence the opposite ulnar nerve block systemically.
  Other Names: dexdor
  Arms: Systemic dexmedetomidine
Drug: Isotonic saline — placebo (saline) is administered perineurally in all but the perineural group.
  Other Names: Placebo
  Arms: High dose Ropivacaine; Placebo; Systemic dexmedetomidine

SUMMARY:
The aim of this trial is to investigate if dexmedetomidine prolongs the duration of an ulnar nerve block. By using healthy volunteers the investigators can perform bilateral ulnar nerve blocks and thereby control for a systemic effect to clarify if the effect is actually peripheral or systemic. The investigators hypothesis is that dexmedetomidine as an adjunct to a local anaesthetic prolongs the duration of a peripheral nerve block by a peripheral mechanism.

DETAILED DESCRIPTION:
Background:

Efficient pain management promoting mobilization and convalescence is essential in an ideal perioperative course. Regional nerve blocks are a central element in postoperative regimes for many patients and it is therefore important that these nerve blocks are both long lasting and efficient. This trial will investigate whether it is possible to optimize the postoperative pain management when adding dexmedetomidine to the local anaesthetic ropivacaine in peripheral nerve blocks.

The prolonging effect of using dexmedetomidine as adjunct in peripheral nerve blocks have been investigated in several studies. However, it remains uncertain whether the effect is mediated by a systemic-, a peripheral- or a combined systemic/peripheral mechanism. In this trial the adjuvating effect of dexmedetomidine will be investigated using an ulnar nerve block.

Method:

The participants will attend two trial days.

On one trial day the volunteers will receive bilateral ulnar nerve blocks. In one arm they will receive the local anaesthetic ropivacaine 4ml 5mg/ml and placebo (saline) and in the other arm ropivacaine 4ml 5mg/ml and dexmedetomidine 100μg. The dexmedetomidine administered perineurally is absorbed and redistributed and will influence the two nerve blocks equally systemically. On the other trial day the participants will receive ropivacaine 4ml 5mg/ml and placebo (saline) and in the other arm ropivacaine 4ml 7.5mg/ml and placebo (saline). The allocation is blinded to volunteer and investigator.

In this setup we therefore have a perineural- and a systemic dexmedetomidine group and also a placebo group , and a group testing if higher doses of local anesthetics will prolong the duration of a nerve block.

The duration of the nerve block will be measured by 3 different tests: pinprick, temperature test (alcohol) and Pain during tonic heat stimulation. All tests are validated within pain research.

ELIGIBILITY:
Inclusion Criteria:

* Participants must understand the protocol fully and sign the written in-formed consent.
* ASA 1-2
* BMI > 18 to < 30
* For fertile women: safe contraceptives for the last month and a nega-tive urin HCG.

Exclusion Criteria:

* Participants unable to cooperate in the trial.
* Participants unable to speak or read Danish
* Allergy to study medication.
* Alcohol consumption >21 units for men and >14 for women per week
* Daily intake of prescription painkillers within the last 4 weeks.
* Over the counter painkillers during the last 48 hours.
* Neuromuscular defects or wounds on the arms or hands preventing test performance.
* Diabetes Mellitus
* 2. degree heart block
* Sick sinus node.
* For fertile women a positive urine HCG

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Difference in duration of sensory nerve block assessed by mechanical discrimination (pinprick) between perineural dexmedetomidine and placebo | 0-36 hours
  Duration of sensory nerve block measured by mechanical discrimination (pinprick) defined as time from block performance (removal of the needle) until the needle feels sharp again.
Difference in duration of sensory nerve block assessed by mechanical discrimination (pinprick) between systemic dexmedetomidine and placebo | 0-36 hours
  Duration of sensory nerve block measured by mechanical discrimination (pinprick) defined as time from block performance (removal of the needle) until the needle feels sharp again.
Difference in duration of sensory nerve block assessed by mechanical discrimination (pinprick) between systemic dexmedetomidine and perineural dexmedetomidine | 0-36 hours
  Duration of sensory nerve block measured by mechanical discrimination (pinprick) defined as time from block performance (removal of the needle) until the needle feels sharp again.

SECONDARY OUTCOMES:
Difference in duration of sensory nerve block assessed by mechanical discrimination (pinprick) between high dose ropivacaine and placebo | 0-36 hours
  Duration of sensory nerve block measured by mechanical discrimination (pinprick) defined as time from block performance (removal of the needle) until the needle feels sharp again.
Difference in duration of sensory nerve block assessed by temperature discrimination between perineural dexmedetomidine and placebo | 0-36 hours
  Duration of sensory nerve block measured by temperature discrimination defined as time from block performance (removal of the needle) until the stimulation with an alcohol swab feels cold again.
Difference in duration of sensory nerve block assessed by temperature discrimination between systemic dexmedetomidine and placebo | 0-36 hours
  Duration of sensory nerve block measured by temperature discrimination defined as time from block performance (removal of the needle) until the stimulation with an alcohol swab feels cold again.
Difference in duration of sensory nerve block assessed by temperature discrimination between systemic dexmedetomidine and perineural dexmedetomidine | 0-36 hours
  Duration of sensory nerve block measured by temperature discrimination defined as time from block performance (removal of the needle) until the stimulation with an alcohol swab feels cold again.
Difference in duration of sensory nerve block assessed by temperature discrimination between high dose ropivacaine and placebo | 0-36 hours
  Duration of sensory nerve block measured by temperature discrimination defined as time from block performance (removal of the needle) until the stimulation with an alcohol swab feels cold again.
Difference in duration of sensory nerve block assessed by pain during tonic heat stimulation between perineural dexmedetomidine and placebo | 0-36 hours
  Duration of sensory nerve block measured by pain during tonic heat stimulation defined as time from block performance (removal of the needle) until a thermode heated to 45C for 30 seconds elicits a painful response again (VAS>0)
Difference in duration of sensory nerve block assessed by pain during tonic heat stimulation between systemic dexmedetomidine and placebo | 0-36 hours
  Duration of sensory nerve block measured by pain during tonic heat stimulation defined as time from block performance (removal of the needle) until a thermode heated to 45C for 30 seconds elicits a painful response again (VAS>0)
Difference in duration of sensory nerve block assessed by pain during tonic heat stimulation between perineural dexmedetomidine and systemic dexmedetomidine | 0-36 hours
  Duration of sensory nerve block measured by pain during tonic heat stimulation defined as time from block performance (removal of the needle) until a thermode heated to 45C for 30 seconds elicits a painful response again (VAS>0)
Difference in duration of sensory nerve block assessed by pain during tonic heat stimulation between high dose ropivacaine and placebo | 0-36 hours
  Duration of sensory nerve block measured by pain during tonic heat stimulation defined as time from block performance (removal of the needle) until a thermode heated to 45C for 30 seconds elicits a painful response again (VAS>0)
Difference in duration of motor nerve block assessed by maximum voluntary isometric contraction between perineural dexmedetomidine and placebo | 0-36 hours
  Duration of motor nerve block measured by maximum voluntary isometric contraction is defined as time from block performance (removal of the needle) until fifth finger abduction maximal voluntary isometric contraction (MVIC) > 75% of baseline value, or the participant indicates return of normal motor funktion.
Difference in duration of motor nerve block assessed by maximum voluntary isometric contraction between systemic dexmedetomidine and placebo | 0-36 hours
  Duration of motor nerve block measured by maximum voluntary isometric contraction is defined as time from block performance (removal of the needle) until fifth finger abduction maximal voluntary isometric contraction (MVIC) > 75% of baseline value, or the participant indicates return of normal motor funktion.
Difference in duration of motor nerve block assessed by maximum voluntary isometric contraction between systemic dexmedetomidine and perineural dexmedetomidine | 0-36 hours
  Duration of motor nerve block meassured by maximum voluntary isometric contraction is defined as time from block performance (removal of the needle) until fifth finger abduction maximal voluntary isometric contraction (MVIC) > 75% of baseline value, or the participant indicates return of normal motor funktion.
Difference in duration of motor nerve block assessed by maximum voluntary isometric contraction between high dose ropivacaine and placebo | 0-36 hours
  Duration of motor nerve block measured by maximum voluntary isometric contraction is defined as time from block performance (removal of the needle) until fifth finger abduction maximal voluntary isometric contraction (MVIC) > 75% of baseline value, or the participant indicates return of normal motor funktion.
Difference in onset of sensory nerve block assessed by mechanical discrimination (pinprick) between perineural dexmedetomidine and placebo | 0-36 hours
  Onset of sensory nerve block assessed by mechanical discrimination (pinprick) is defined as time from block performance (removal of the needle) until the needle stops feeling sharp.
Difference in onset of sensory nerve block assessed by mechanical discrimination (pinprick) between systemic dexmedetomidine and placebo | 0-36 hours
  Onset of sensory nerve block assessed by mechanical discrimination (pinprick) is defined as time from block performance (removal of the needle) until the needle stops feeling sharp.
Difference in onset of sensory nerve block assessed by mechanical discrimination (pinprick) between perineural dexmedetomidine and systemic dexmedetomidine | 0-36 hours
  Onset of sensory nerve block assessed by mechanical discrimination (pinprick) is defined as time from block performance (removal of the needle) until the needle stops feeling sharp.
Difference in onset of sensory nerve block assessed by mechanical discrimination (pinprick) between high dose ropivacaine and placebo | 0-36 hours
  Onset of sensory nerve block assessed by mechanical discrimination (pinprick) is defined as time from block performance (removal of the needle) until the needle stops feeling sharp.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob H Andersen, M.D., Principal Investigator — Department of Anesthesiology, Zealand University Hospital
Locations (1):
- Department of Anesthesiology Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Andersen JH, Jaeger P, Grevstad U, Estrup S, Geisler A, Vilhelmsen F, Dahl JB, Laier GH, Ilfeld BM, Mathiesen O. Systemic dexmedetomidine is not as efficient as perineural dexmedetomidine in prolonging an ulnar nerve block. Reg Anesth Pain Med. 2019 Mar;44(3):333-340. doi: 10.1136/rapm-2018-100089. Epub 2019 Jan 23. PMID 30679332